CLINICAL TRIAL: NCT03043014
Title: Cervical Preparation of Abortions Under Paracervical Block in the First Trimester: A Randomized Clinical Trial
Brief Title: Cervical Preparation of Abortions Under Paracervical Block in the First Trimester:
Acronym: BPCEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-35
Record Dates: First submitted 2017-01-25; First posted 2017-02-03 (Estimated); Last update posted 2022-11-16 (Actual); Status verified 2019-11

CONDITIONS: Surgical Abortion

STUDY DESIGN:
Intervention Model Description: The women will be randomized into two groups: Mifépristone group and Misoprostol group. The main endpoint will be the per-operating pain. The other endpoints are the pre and post-operative pain, the complications (cervical tearing, uterine perforation, hemorrhage requiring the use of blood products or an hemostatic intervention), the surgical time necessary to terminate the pregnancy, the side-effects of the drugs. The amount of per-operating bleeding and the duration of the intervention . We assume that the use of Mifepristone in the cervical preparation of the surgical abortion under LA would reduce the per-operating pain. The number of patients required is 55 in each arm.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mifépristone group (Experimental)
  Interventions: Drug: Mifépristone versus Misoprostol
- misoprostol group (Active Comparator)
  Interventions: Drug: Mifépristone versus Misoprostol

INTERVENTIONS:
Drug: Mifépristone versus Misoprostol — The women will be randomized into two groups: Mifépristone group and Misoprostol group. The main endpoint will be the per-operating pain. The other endpoints are the pre and post-operative pain, the complications (cervical tearing, uterine perforation, hemorrhage requiring the use of blood products or an hemostatic intervention), the surgical time necessary to terminate the pregnancy, the side-effects of the drugs. The amount of per-operating bleeding and the duration of the intervention . The investigators assume that the use of Mifepristone in the cervical preparation of the surgical abortion under LA would reduce the per-operating pain. The number of patients required is 55 in each arm.

SUMMARY:
Surgical abortion is one of the most frequently surgery of women in the world. 43 millions are annually performed in the world.

90% of the abortions are performed during the first trimester of pregnancy before 13 weeks. Legal surgical abortion during the first trimester of pregnancy is a low risk intervention with a mortality rate lower than 1/100 000 abortions, with a risk of complications from 0.3 % to 3.4 %.

DETAILED DESCRIPTION:
Surgical abortion is one of the most frequently surgery of women in the world. 43 millions are annually performed in the world.

Legal surgical abortion during the first trimester of pregnancy is a low risk intervention with a mortality rate lower than 1/100 000 abortions, with a risk of complications from 0.3 % to 3.4 %. In France, about 75 % of the surgical abortions are performed under general anesthesia (GA). Nevertheless, the risk of complications is higher under GA. The risk of death is more important (0,58 for 100 000) with GA. GA increases by a factor 1,7 the risk of bleeding, 2,2 the risk of uterine perforation, 8,2 the risk of intra-abdominal bleeding, 2,9 the risk of cervical tearing, and 5 the risk of transfusion. The difficulty of pain control under local anesthetia (LA) explains this method is less choosen by the women. Indeed, a lot of women consider the surgical abortion under LA extremely uncomfortable. The paracervical block for the abortion under LA in the first trimester demonstrated its efficiency in the reduction of the per-operating pain whatever the term of the pregnancy compared with the absence of anesthesia. The cervical preparation demonstrated benefits in term of cervical dilation, per-operating bleeding, and complications incidence. The misoprostol and the mifepristone are 2 molecules recommended for the cervical preparation on the first trimester

ELIGIBILITY:
Inclusion Criteria:

aged 18 or over with a single intra uterine pregnancy whose term is between 6 and 14 weeks the day of the abortion estimated by ultrasound by a measurement of the cranio-caudal length between 5 and 84 millimeters surgical abortion under local anesthesia informed written consent

Exclusion Criteria:

minor multiple pregnancy Uterine malformation coagulation disorder defined by biological parameters (TP<70%, TCA patient / control ratio < 1.20) Allergy or hypersensitivity to any of the active substance or to any of the excipients Contraindication to mifepristone chronic renal insufficiency severe asthma uncontrolled by treatment hereditary porphyria allergy to the active substance or to any of the excipients; not affiliated to the social security system; no informed consent. Suspicion of ectopic pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
per operative pain | 20 minutes
  It is carried out using a numerical scale rated from 0 to 10 (0 absence of pain, 10 maximum of pains felt).
Anxiety | 48 hours
  STAI anxiety questionnaire;it is a self-questionnaire, developed by Spielberger (Spielberger, 1983) and validated in French (Gauthier & Bouchard, 1993). It consists of 20 questions, assessing the usual emotional state of the subject. A score is calculated, a high score indicating the presence of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital de la conception Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamdaoui N, Cardinale C, Fabre C, Baumstarck K, Agostini A. Pain Associated With Cervical Priming for First-Trimester Surgical Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jun 1;137(6):1055-1060. doi: 10.1097/AOG.0000000000004376. PMID 33957651